CLINICAL TRIAL: NCT00170053
Title: Randomized Trial of Thymoglobulin Induction, Initial Tacrolimus, and Mycophenolate Mofetil Therapy With Steroid Avoidance in Primary Kidney Transplant Recipients Followed by Continued Tacrolimus/Mycophenolate Mofetil Therapy vs. Sirolimus/ Mycophenolate Mofetil Therapy
Brief Title: Comparison of Sirolimus to Tacrolimus for Long Term Therapy in Kidney Transplant With no Steroids
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Genzyme, a Sanofi Company (Industry); Raymond Heilman (Unknown)
Responsible Party: Thomas A. Gonwa, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 37-05; Wyeth 0468H-101898
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Kidney Diseases
Keywords: Kidney Transplantation
MeSH Terms: conditions — Kidney Diseases | interventions — Sirolimus

INTERVENTIONS:
Drug: Sirolimus — 10 mg oral loading dose followed by 5 mg/day. Measure Sirolimus level weekly and adjust to level of 10-15 ng/ml.

SUMMARY:
Kidney transplant patients will be treated with Thymoglobulin (5 days), tacrolimus (Prograf), and mycophenolate mofetil (Cellcept) from the time of transplant. They will only receive steroids for 4 days and no prednisone after that. At 1 month, they will have a kidney biopsy and if it is ok, patients will be treated long term with either continued tacrolimus/mycophenolate mofetil or be switched to sirolimus (Rapamune)/mycophenolate mofetil. This will be done randomly in a manner similar to flipping a coin. The investigators are trying to determine if after the initial therapy patients can stay off steroids long term and get better kidney function if they are treated with sirolimus compared to tacrolimus. Patients will be followed for 3 years and will repeat kidney biopsies at 1 and 2 years after transplant.

DETAILED DESCRIPTION:
Abstract:

Corticosteroids have been a mainstay of immunosuppression for kidney transplantation, but they are associated with significant toxicity after long-term use. Recent studies have concluded that steroid avoidance is safe and effective when combined with modern immunosuppressive maintenance therapy in low risk kidney transplant recipients. These studies have included antilymphocyte induction therapy with either an anti IL-2 receptor antibody, or an antithymocyte globulin, such as rabbit polyclonal antithymocyte globulin (Thymoglobulin). Mayo Clinic Scottsdale has adopted Thymoglobulin induction, tacrolimus, and mycophenolate mofetil with rapid steroid taper as their standard immunosuppressive therapy in low risk patients. Mayo Clinic Jacksonville is also utilizing this protocol. Together, both sites have utilized this approach in 64 patients. Recent improvements in immunosuppressive regimens have decreased acute rejection in kidney transplant recipients and increased one-year graft survival to nearly 90%. However, long-term graft survival has changed little with 30% of grafts being lost to ''chronic allograft nephropathy'' (CAN) in the first five years after transplantation. A recent paper highlighted this dilemma and demonstrated that a major cause of late CAN was chronic exposure to the nephrotoxic effects of calcineurin inhibitors (CNI) tacrolimus and cyclosporine and possibly cytomegalovirus infection. In this study, we will focus on the role of CNI in CAN. We propose a prospective, randomized, non-blinded trial of Thymoglobulin induction with rapid steroid elimination accompanied by tacrolimus (TAC) and mycophenolate mofetil (MMF) maintenance therapy. Patients are to be randomized at 1 month post-operatively to either remain on TAC/MMF or switch to SRL/MMF. The primary endpoint will be renal function at 1-year post-transplant. Secondary endpoints will include renal function at 2 years post-transplant, histology seen on protocol biopsies at 1 and 2 years post-transplant, incidence of biopsy proven rejection at 12 months, patient survival, graft survival, proportion of patients steroid free at 12 months, infectious complications, bone mineral density analysis, incidence of hyperlipidemia, and the incidence of new onset post-transplant diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Primary deceased or living donor renal transplant recipients
2. Re-transplant recipients for which the first kidney transplant was lost for technical reasons with no sensitization (panel-reactive antibody [PRA] < 20%) or 1st lost due to recurrent disease, that is not steroid responsive.
3. Age > 18
4. Negative pregnancy test if female and of childbearing age. In addition, females of childbearing age must agree to use effective contraception for the duration of the study.
5. Patient must sign informed consent prior to transplant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2005-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Renal function | 1 year

SECONDARY OUTCOMES:
Renal function | 2 years
Transplant biopsy histology | 2 years
Patient and graft survival | 2years
Acute rejection rate | 1 month
Number of patients steroid free | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A. Gonwa, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States